CLINICAL TRIAL: NCT03759171
Title: Music-instruction Intervention for Treatment of Post-traumatic Stress Disorder: A Randomized Pilot Study
Brief Title: Music-instruction Intervention for Treatment of Post-traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Milwaukee VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Liliana Pezzin, Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO00019269
Record Dates: First submitted 2018-11-16; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Stress Disorders, Post-Traumatic; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: Delayed entry, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Entry Group (Experimental): Following the baseline interview, veterans randomized to the immediate entry group directly engaged in the Guitars for Vets Intervention and were interviewed at the end of the intervention period, roughly 6 weeks later. The intervention content and duration (6 weeks) was the same across both groups.
  Interventions: Other: Guitars for Vets Intervention
- Delayed Entry Group (Experimental): Those randomized to the delayed entry group had their baseline interview repeated at the end of the delayed entry period (4 weeks) prior to receiving the 6-week Guitars for Vets Intervention as well as after intervention completion. The intervention content and duration (6 weeks) was the same across both groups.
  Interventions: Other: Guitars for Vets Intervention

INTERVENTIONS:
Other: Guitars for Vets Intervention — This was an active intervention providing veterans with an acoustic guitar, guitar pick, tuning instruments, a music book, practice CDs, and individual and group sessions of music instruction during a 6-week intervention period. Six tailored 1-hour individual guitar instruction sessions were scheduled (1 session per week). In addition to the 6 tailored individual lessons, the intervention provided 3 group sessions. Veterans were given a guitar that they could keep upon completion of the program. The same instructor was assigned to a subject for the duration of the study, and group sessions were supervised by the Education Director of Guitars for Vets.

SUMMARY:
The purpose of this study was to examine the feasibility and potential effectiveness of an active, music-instruction intervention in improving psychological health and social functioning among Veterans suffering from moderate to severe Post-traumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
The study was designed as a prospective, delayed-entry randomized pilot trial. Regression-adjusted difference in means were used to examine the intervention's effectiveness with respect to PTSD symptomatology (primary outcome) as well as depression, perceptions of cognitive failures, social functioning and isolation, and health-related quality of life (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Veterans who (i) had at least one visit for mental health treatment in the prior six months with a primary diagnosis of PTSD (ICD9CM 309.81-83) and (ii) exhibited moderate to severe PTSD symptoms at the time of enrollment (Posttraumatic Stress Disorder Checklist >=50)

Exclusion Criteria:

* Veterans who were currently participating in an intense psychotherapy program (residential or outpatient)
* Veterans who were already receiving guitar lessons from a Guitars for Vets volunteer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder (PTSD) Symptoms | 6 weeks
  Post-Traumatic Stress Disorder (PTSD) symptoms as measured by the PTSD Checklist Civilian (PCLC), a self-report scale that measures PTSD presence and severity. The 17 items correspond to Diagnostic and Statistical Manual DSM-IV symptoms of PTSD. The level of distress produced by each symptom is rated from 1 (not at all) to 5 (extremely). A score >50 on this measure is considered clinically significant (maximum score = 85).

SECONDARY OUTCOMES:
Depression | 6 weeks
  Depression was assessed using the Beck Depression Inventory-II (BDI-II), a 21-item self-report scale measuring the presence and severity of depressive symptoms over the two weeks preceding test administration. Each answer ranges in score from 0-3. Total scores indicate minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63; maximum = 63) levels of reported depression.
Perceptions of Cognitive Failures | 6 weeks
  The Cognitive Failures Questionnaire (CFQ) was used as a self-reported measure of everyday cognitive lapses for perception, memory, and motor function, such as forgetting appointments or having word finding difficulty. Total scores range from 0 to 100 with higher numbers indicating worse outcomes.
Social Functioning | 6 weeks
  The University of California, Los Angeles (UCLA) Loneliness Scale was administered to assess subjective feelings of social isolation. This is a 20-item scale summed to give a total score ranging from 0-60 with higher numbers indicating worse outcomes.
Health-Related Quality of Life | 6 weeks
  The European Quality of Life (EuroQoL) Scale, a validated preference-based scale for which population norms are available in the US and elsewhere, was used as the global evaluation of veteran's health-related quality of life. The 5-item EuroQoL measure combines data on activity restrictions (ADL, IADL limitations), limitations in participation (usual major activity and other social activities) and self- perceived health status (excellent, good, fair or poor) to measure one's overall satisfaction with health and well-being. Scores range from -0.594 to 1.000, higher values represent better outcomes.

IPD SHARING:
Plan to Share IPD: No